CLINICAL TRIAL: NCT05806723
Title: Effects of High Intensity Statin Therapy on Steroid Hormones and Vitamin D in Type 2 Diabetic Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital La Rabta (Other)
Responsible Party: Principal Investigator, Melika Chihaoui, Professor, University Tunis El Manar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLaRabta22021
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2; Dyslipidemia Associated With Type II Diabetes Mellitus; Statin Adverse Reaction; Hypogonadism, Male; Adrenal Insufficiency; Vitamin D Deficiency
Keywords: type 2 diabetes; statin; testosterone; cortisol; vitamin D; DHEAS
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Eunuchism; Adrenal Insufficiency; Vitamin D Deficiency | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- type 2 diabetic patients at high cardio vascular risk (Experimental): atorvastatin 40 mg a day for six months
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — daily drug intake during six months

SUMMARY:
The aim of the study was to assess the effect of high intensity statin therapy on testicular and adrenal steroids and vitamin D levels in type 2 diabetes males.It is a prospective study, conducted between march 2021 and July 2022, including 60 men with type 2 diabetes, aged 40 - 65 years, statin-free, and in whom a treatment with high intensity statin was indicated. The patients had two visits, before and six months after a daily intake of 40 mg of atorvastatin. During each visit, they underwent a clinical examination including the Androgen Deficiency in the Aging Male (ADAM) questionnaire and a fasting blood sample was collected for biological and hormonal measurements.

DETAILED DESCRIPTION:
Study design and setting It is a prospective study carried out at the department of Endocrinology of the University Hospital La Rabta, Tunis, between March 2021 and July 2022. The protocol was approved by La Rabta University Hospital local ethics committee.

Subjects Inclusion criteria were male subjects, aged between 40 and 65 years, with T2D, naive to statin and in whom a high intensity statin therapy was indicated according to the recommendations of the American Diabetes Association 2021 i.e in secondary cardio-vascular prevention or in primary prevention if the patient was aged more than 50 years or if other atherosclerotic cardiovascular disease risk factors were associated.

All patients gave an informed written consent to participate in the study. Exclusion criteria were the use within the last six months of drugs interfering with steroidogenesis (androgens, anti-androgens, Gn-RH analogues, corticosteroids, antiepileptics, barbiturates or other enzyme inducer or inhibitor); history of endocrinopathy (hypogonadism, testicular tumor, pituitary insufficiency, adrenal insufficiency, uncontrolled hypothyroidism); history of severe systemic disease (hepatic insufficiency, cirrhosis, alcoholism, severe or moderate renal insufficiency, symptomatic heart failure, chronic inflammatory disease); myocardial infarction or stroke within the last six months; statin intolerance; withdrawal of consent; loss to follow-up; poor compliance with treatment.

The number of subjects required for the study was calculated. When considering alpha= 0.05, beta= 0.10, and a magnitude of difference in testosterone levels of 0.59 ng/ml according to Dobs AS et al. study with an estimated common standard deviation of 1.0, the number of subjects required is estimated to be 50.

Protocol and data collection Visit 1: inclusion visit. The subjects were included and signed an informed consent to participate in the study. Visits 1 and 2 were performed on the same day in fasting patients.

Visit 2:

Clinical data were determined: age; habits; history; ongoing treatment; signs of adrenal insufficiency (weight loss, anorexia, asthenia, dizziness on standing, signs of hypoglycemia); signs of hypogonadism (decreased libido, presence or absence of nocturnal erections); number of sexual intercourses per month. Patients responded to the androgen deficiency in the aging male questionnaire (ADAM) translated to Tunisian dialect by four physicians from the same department.

Patients underwent a physical examination: measure of weight, height, and lying and standing blood pressure, presence of melanoderma, gynecomastia or myalgia.

A blood sample was collected between 8 a.m. and 9 a.m., after 12 hours of fasting, for the measurement of glucose, HbA1c, total cholesterol, triglycerides, high density lipoprotein cholesterol (HDLc), creatinine, sodium, potassium, transaminases (alanine aminotransferase (ALT) and aspartate aminotransferase (AST)), creatine phosphokinase (CPK), calcium, phosphate, albumin, total testosterone, sex hormone binding globulin (SHBG), estradiol, follicle stimulating hormone (FSH), luteinizing hormone (LH), cortisol, DHEAS (dehydroepiandrosterone sulfate), parathormone (PTH), and 25-hydroxy vitamin D. Blood samples were frozen at -20°c at the laboratory until hormonal measurements.

Treatment with 40 mg atorvastatin a day was initiated in all patients.

Visit 3: after six months of treatment:

The clinical and paraclinical parameters determined at visit 1 were determined again. The dose and the compliance of statin intake were evaluated by Girerd questionnaire. The occurrence of clinical adverse events of statin such as myalgia, arthralgia, digestive symptoms was recorded.

ELIGIBILITY:
Inclusion Criteria:

* male subjects
* aged between 40 and 65 years
* Type 2 diabetes
* naive to statin
* patients in whom a high intensity statin therapy was indicated according to the recommendations of the American Diabetes Association 2021 i.e in secondary cardio-vascular prevention or in primary prevention if the patient was aged more than 50 years or if other atherosclerotic cardiovascular disease risk factors were associated.

Exclusion Criteria:

* the use within the last six months of drugs interfering with steroidogenesis (androgens, anti-androgens, Gn-RH analogues, corticosteroids, antiepileptics, barbiturates or other enzyme inducer or inhibitor)
* history of endocrinopathy (hypogonadism, testicular tumor, pituitary insufficiency, adrenal insufficiency, uncontrolled hypothyroidism)
* history of severe systemic disease (hepatic insufficiency, cirrhosis, alcoholism, severe or moderate renal insufficiency, symptomatic heart failure, chronic inflammatory disease)
* myocardial infarction or stroke within the last six months
* statin intolerance
* withdrawal of consent
* loss to follow-up
* poor compliance with treatment.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male gender
Enrollment: 104 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
change in testosterone level after atorvastatin treatment | six months
  decrease in testosterone level

SECONDARY OUTCOMES:
change in cortisol level after atorvastatin treatment | six months
  decrease in cortisol
change in DHEAS levels after atorvastatin treatment | six months
  decrease in DHEAS

OTHER OUTCOMES:
change in vitamin D level after atorvastatin treatment | six months
  decrease in vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Melika Chihaoui, Professor, Principal Investigator — La rabta hospital
Locations (1):
- University Hospital La Rabta, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after the publication
Access Criteria: on request

REFERENCES:
- [Derived] Chihaoui M, Terzi A, Hammami B, Oueslati I, Khessairi N, Chaker F, Yazidi M, Feki M. Effects of high-intensity statin therapy on steroid hormones and vitamin D in type 2 diabetic men: A prospective self-controlled study. Lipids. 2024 Sep;59(5):135-144. doi: 10.1002/lipd.12399. Epub 2024 May 20. PMID 38764377